CLINICAL TRIAL: NCT07397988
Title: Feasibility Study for Logistics and Data Stability of Continuous Temperature Monitoring Using a Wearable Device With a Continuous Core Temperature Reference Method
Brief Title: Feasibility of Wearable-Based Continuous Temperature Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: am25Eckstein4
Record Dates: First submitted 2026-01-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Temperature Change, Body
Keywords: Continuous temperature monitoring; Wearable devices; Feasibility study; Ingestible temperature capsule; Real-world monitoring
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ingestible temperature capsule
  Interventions: Device: Continuous Temperature Monitoring

INTERVENTIONS:
Device: Continuous Temperature Monitoring — Participants wear investigational temperature sensors and ingest a core temperature capsule continuous data collection

SUMMARY:
The aim of this study is to evaluate the feasibility of collecting synchronised continuous temperature data using wearable devices and a continuous core temperature reference under real-world conditions. The study focuses on workflow execution, data continuity, secure retrieval, and time-alignment without diagnostic or therapeutic intent.

DETAILED DESCRIPTION:
Continuous temperature monitoring in real-world and free-living settings is operationally challenging due to intermittent standard measurements and context-dependent variability. This limits the ability to evaluate the integrity and stability of continuous temperature time-series and to test end-to-end data collection workflows.

This feasibility study is conducted to determine whether synchronised continuous temperature data from wearable devices and an ingestible core temperature reference can be collected, time-aligned, and retrieved reliably with acceptable participant and staff burden. The study generates feasibility evidence on workflow performance and data stability to inform the design of a subsequent confirmatory clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any project-specific procedures.
* Age 18 years or older at enrolment.
* Able and willing to comply with project procedures, including capsule ingestion, continuous wearable use for around 48 hours, and adherence to study instructions.
* Able to swallow the ingestible temperature capsule without difficulty.
* No contraindication to ingestible thermometry as assessed by the investigator.

Exclusion Criteria:

General:

* Body weight < 36 kg.
* Women who are pregnant.
* Participation in another clinical investigation involving an investigational medicinal product or medical device within the 30 days preceding enrolment or previous enrolment in the current project.
* Enrolment of the Principal Investigator, project staff, their family members, employees, or other dependent persons.
* Inability to provide valid informed consent or significant language barrier preventing adequate understanding of procedures.

Implants & MRI:

* Presence of any active Implantable Medical Device (AIMD), including Pacemakers, Implantable Cardioverter Defibrillators (ICDs), Deep Brain Stimulation (DBS) devices, or Left Ventricular Assist Devices (LVADs).
* Requirement for MRI scanning during the seven days following the capsule intake.

Cognitive/Physical Status:

* Unconscious patients (prior to ingestion).
* Patients with special needs or disabilities preventing safe autonomous swallowing.

Gastrointestinal:

* Known history of dysphagia or gag reflex troubles.
* Previous gastrointestinal surgery resulting in bowel stenosis.
* Current or planned surgical procedures on the GI tract (esophagus, stomach, intestines).
* Zenker's diverticulum or felinization of the esophagus.
* Risk or history of intestinal obstruction, strictures, or diverticula.
* Hypomotility disorders (e.g., ileus).
* Inflammatory Bowel Diseases including Crohn's disease or Ulcerative Colitis.

Dermatological Exclusions (Rheo Vital+ Performance)

* Dermatological conditions, wounds, tattoos, oedema, inflammation, active venous access, or other impairments at the medial upper arm or axillary region that could interfere with correct placement or functioning of the wearable device.
* Excessive hair or concurrent devices that hinder correct sensor placement.
* Known allergy to plastics or latex.

Temperature Management:

* Active external heating or cooling (e.g., cooling blankets).
* Note: Use of pharmacological antipyretics (oral/IV) is permitted.

Further Medical Conditions:

* Currently existing acute back pain.
* Symptomatic herniated disc.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult participants (≥18 years) capable of providing informed consent and willing to comply with the project procedures, including ingestion of the capsule and continuous wearing of two wearable devices for around 48 hours until capsule excretion under free-living conditions.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Paired Continuous Temperature Data Completeness | Baseline to 48 hours
  Participant-level paired data completeness (%) over the planned monitoring period, defined as the proportion of monitoring minutes with usable and time-aligned temperature data from both the wearable device(s) and the ingestible capsule.

SECONDARY OUTCOMES:
Recruitment and Retention Feasibility | Baseline to 48 hours
  Proportion of eligible participants enrolled among those approached and proportion of enrolled participants completing the planned monitoring period.
Data continuity (wearable data) | Baseline to 48 hours
  Percent expected time with usable wearable data
Data continuity (wearable data) | Baseline to 48 hours
  Categorised reasons for missing/invalid data
Data continuity (capsule data) | Baseline to 48 hours
  frequency/duration of gaps
Data continuity (capsule data) | Baseline to 48 hours
  Percent expected time with usable capsule data
Data continuity (capsule data) | Baseline to 48 hours
  Categorised reasons for missing/invalid data
Time-alignment success between wearable and capsule streams | Baseline to 48 hours
  Success rate of time synchronisation
Time-alignment success between wearable and capsule streams | Baseline to 48 hours
  Distribution of residual alignment error after the defined alignment procedure (reported descriptively).
Data retrieval workflow | Baseline to 48 hours
  Success rate of secure data retrieval/transfer
Data retrieval workflow | Baseline to 48 hours
  Number of troubleshooting events
Data retrieval workflow | Baseline to 48 hours
  Time spent per participant
Tolerability Questionnair | Baseline to 48 hours
  Participant-reported tolerability and wear adherence assessed by a questionnaire
Tolerability: skin discomfort | Baseline to 48 hours
  Incidence and nature of wearable skin discomfort
Tolerability: GI discomfort | Baseline to 48 hours
  Capsule-related GI discomfort/delayed excretion (descriptive)
Observed temperature trajectories | Baseline to 48 hours
  Descriptive summaries of temperature time courses; whether transient elevations >38.0°C were captured
Baseline factors considered (descriptive stratification only) | Baseline to 48 hours
  Age and sex will be explored descriptively as potential drivers of data quality metrics
Baseline factors considered (descriptive stratification only) | Baseline to 48 hours
  Age and sex will be explored descriptively as potential drivers of observed temperature dynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, Prof. MD, Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland